CLINICAL TRIAL: NCT05707013
Title: Comparing Efficacy Between Traditionally Fabricated Foot Orthotics and the HP Arize 3D Printed Foot Orthotics
Brief Title: HP Arize 3D Orthotics for Planar Fasciitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Midlands (Other)
Collaborators: Hewlett-Packard (HP) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1876792
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Plantar Fascitis
Keywords: orthotics

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive traditionally fabricated orthotics or HP Arize 3D-printed orthotics for treatment of plantar fasciitis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HP Arize 3D-Printed Orthotics (Experimental): Patients will receive the HP Arize 3D-printed orthotics for treatment of plantar fasciitis.
  Interventions: Device: HP Arize 3D-Printed Orthotics
- Traditional Orthotics (Active Comparator): Patients will receive traditionally fabricated orthotics for treatment of plantar fasciitis.
  Interventions: Device: Traditional Orthotics

INTERVENTIONS:
Device: HP Arize 3D-Printed Orthotics — Custom 3D-printed orthotics manufactured by HP.
  Arms: HP Arize 3D-Printed Orthotics
Device: Traditional Orthotics — Traditionally fabricated custom orthotics manufactured by a local supplier.
  Arms: Traditional Orthotics

SUMMARY:
Currently 77% of Americans experience foot pain, of which a large portion can be attributed to plantar fasciitis.

The Arize Orthotic solution, developed in collaboration with podiatrists and leading industry experts, is a new digital solution that helps podiatrists create custom foot orthoses tailored to the patient, quickly, easily, accurately, and reliably. This pilot study will evaluate the effectiveness and clinical benefit of 3D printed foot orthotics compared to traditionally fabricated custom-made orthotics and assess compliance and patient satisfaction in patients with plantar fasciitis.

DETAILED DESCRIPTION:
Currently 77% of Americans experience foot pain, of which a large portion can be attributed to plantar fasciitis. Approximately half of the people with foot pain do not consult a doctor due to cost, convenience, or insurance reasons. To this end, HP will implement an end-to-end system to provide 3D-printed custom orthotic inserts to patients in a fast and efficient manner via their podiatrist.

The Arize Orthotic solution developed in collaboration with podiatrists and leading industry experts, is a new digital solution that helps podiatrists create custom foot orthoses tailored to the patient, quickly, easily, accurately, and reliably. The Arize Orthotic Solution leverages HP 3D Printing technology and aims to further HP's mission to create technology that makes life better for everyone, everywhere.

This pilot study will evaluate the effectiveness and clinical benefit of 3D printed foot orthotics compared to traditionally fabricated custom-made orthotics and assess compliance and patient satisfaction in patients with plantar fasciitis.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosis of plantar fasciitis
* Access to methods of electronic communication (i.e., email)

Exclusion Criteria:

* Previously prescribed and/or used orthotic inserts
* Requires additional bracing of the lower leg
* Diagnosis of neuropathy, acute fracture, or stress fracture
* Pregnant women
* Non-English speakers
* Medicare patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient-reported compliance and satisfaction with orthotics. | 8 weeks
  Patient-reported compliance with traditionally fabricated or 3D-printed orthotics will be assessed at 4 weeks and 8 weeks post-initiation of orthotic wearing via a study-specific survey. This survey includes questions related to how often the patient wore their orthotics, the ease of the process, and fit and feel of the orthotics, and any experienced side effects. This survey was developed by the research team and includes subjective responses to questions; there is no score associated with this assessment.

SECONDARY OUTCOMES:
Patient-reported secondary site pain following implementation of orthotics. | 8 weeks
  Patient-reported secondary site pain for patients wearing either traditionally fabricated or 3D-printed orthotics will be assessed at the time of consent, 4 weeks, and 8 weeks post-initiation of orthotic wearing via a study-specific survey. This survey asks patients to provide a pain score and function score for 11 locations on the body. Scores range from 0 to 100, with 0 being no pain or no limitation to physical function, and 100 being the worst pain possible or complete limitation to physical function.

CONTACTS AND LOCATIONS:
Locations (1):
- Prisma Health - Midlands, Lexington, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No